CLINICAL TRIAL: NCT00434759
Title: Evaluation of the Efficacy, Mechanisms of Change and Efficiency of a Stepped-care Program With a Computer-based Self-help Module and Minimal Therapist Contact in Comparison to a Standard Cognitive Therapy for Patients With Social Phobia
Brief Title: Social Phobia Intervention Study of Mannheim
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SP-32000
Record Dates: First submitted 2007-02-09; First posted 2007-02-13 (Estimated); Results first posted 2012-11-28 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2012-10

CONDITIONS: Social Phobia
Keywords: randomized controlled trial; stepped-care program; cognitive therapy of social phobia according to D.M. Clark
MeSH Terms: conditions — Phobia, Social | interventions — Cognitive Behavioral Therapy; Water Wells

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SCP (Active Comparator): SCP is a stepped-care program with a self-help module with minimal therapist contact (8 sessions) as first step, followed by therapist-guided intervention depending on status of remission (8 sessions up to a maximum of 16 sessions).
  Interventions: Behavioral: stepped care program based on cognitive therapy
- ST (Active Comparator): A standard therapy which means a therapist-guided intervention with 16 sessions face-to-face therapy.
  Interventions: Behavioral: cognitive therapy

INTERVENTIONS:
Behavioral: cognitive therapy — changing safety behaviors, self-focused attention, and automatic negative thoughts in anxiety-provoking situations via cognitive techniques, for example role plays and behavioral experiments
  Other Names: cognitive therapy of social phobia according to D.M. Clark
  Arms: ST
Behavioral: stepped care program based on cognitive therapy — starting with a digital-video-disk-based (DVD-based) self-help module (8 Sessions) followed by face-to-face-therapy including 8 or 16 sessions depending on remission status; including: changing safety behaviors, self-focused attention, and automatic negative thoughts in anxiety-provoking situations via cognitive techniques, for example role plays and behavioral experiments
  Other Names: based on cognitive therapy for social phobie by Clark & Wells (1995)
  Arms: SCP

SUMMARY:
Primary objective:

The purpose of this study is to examine efficacy and efficiency of a Stepped Care Program (SCP) for patients with Social Phobia in comparison to the standard cognitive therapy for Social Phobia according to D.M. Clark.

Secondary objective:

Further, it is intended to identify mechanisms of change which mediate treatment outcome and to identify differential predictors for therapy success for the two treatment conditions.

DETAILED DESCRIPTION:
With prevalence rates (lifetime) up to 13% in western countries, Social Phobia is one of the most frequent mental disorders. Main objective of this clinical trial is the evaluation of the efficacy and efficiency of a stepped care program for patients with Social Phobia (SCP) as compared to a standard therapy (ST) for patients with social phobia. Both interventions are based on the cognitive therapy according to D.M. Clark.

The SCP starts with a 8-sessions self-help-module with minimal therapist contact via email. Patients who do not reach remission after this first step, enter step 2 which consists of 8 therapy sessions guided by a therapist. If patients are not remitted after that, they receive another 8 sessions of therapist-guided cognitive treatment in step 3. So the SCP contains 8, 16 or 24 sessions of therapy - depending on remission status of the patient. In contrast to that, the ST comprises 16 sessions of therapist-guided intervention.

The diagnostic status of the patients is assessed by blinded clinician raters before treatment, after every eighth therapy session, and at 5 follow-up timepoints in order to examine the stability of treatment effects (3, 6, 9, 12 and 30 months after the end of therapy). Besides efficacy and efficiency of the SCP vs. ST, mechanisms of change and differential predictors for therapy outcome will be investigated.

Hypotheses: We expect that

1. the SCP is significantly more effective than the ST.
2. the SCP is significantly more efficient than the ST.
3. the results referring to the efficacy will be stable up to 30 months after the end of treatment(Follow Up Phase).
4. the SCP will cause less primary and secondary costs than the ST.
5. successful therapy leads to an improvement in the following areas:

   * reduction of biased information processing,
   * reduction of negative thoughts, subjective anxiety, safety behaviors, self-focused attention and autonomic arousal in anxiety-provoking situations,
   * amelioration of verbal and non-verbal social competence in anxiety- provoking situations.

As mediators of change, the factors maintaining social anxiety according to the model of Social Phobia by Clark and Wells (1995) will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Social Phobia according to the criteria of the Diagnostic and Statistical Manual of Mental Disorders IV (DSM-IV)
* Duration of the disorder at least 1 year
* Severity of symptomatology according to at least one of two self-report measures for social anxiety above Cut-Off: Social Interaction Anxiety Scale (SIAS: value of 26 or more) and / or Social Phobia Scale (SPS: value of 17 or more)
* Age: 18-60
* Written Informed Consent

Exclusion Criteria:

* Social Phobia is not the main diagnosis
* Mental Retardation
* Lifetime Diagnoses: Schizophreniform Disorder, Bipolar Affective Disorder
* Acute Diagnoses: severe Major Depression Episode, severe Anorexia Nervosa, Substance-, Drug - or Alcohol-Dependence, life-threatening suicidal crisis
* Psychotropic medication (except stable treatment with antidepressant since 3 months before study start: medication and dosage has to be stable during the entire study duration)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 89 (Actual)
Dates: Start 2006-09; Primary Completion 2009-05 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Bohus, MD, Study Director — Central Institute of Mental Health in Mannheim
Locations (1):
- Central Institute of Mental Health, Mannheim, Baden-Wurttemberg, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Stepped Care Program: stepped-care program with self-help module with minimal therapist contact as first step, followed by therapist-guided intervention depending on status of remission
- Standardtherapy: standard therapy (therapist-guided intervention only)
Period: Overall Study
Arm/Group | Stepped Care Program | Standardtherapy
Started | 46 | 43
Completed | 22 | 38
Not Completed | 24 | 5
Not completed — Lack of Efficacy | 5 | 4
Not completed — Withdrawal by Subject | 17 | 1
Not completed — family affairs | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stepped Care Program | Standardtherapy | Total
Number analyzed (Participants) | 46 | 43 | 89
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 43 | 89
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 37.26 (10.47) | 38.47 (10.26) | 37.84 (10.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 24 | 48
  Male | 22 | 19 | 41
Region of Enrollment [Number; unit: participants]
  Germany | 46 | 43 | 89

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Social Interaction Anxiety Scale (SIAS)
Description: This scale measures interaction anxiety on a 5-point scale (range of scores is 0-4); the number of items is 20; the total minimum for all 20 items is 0 and the total maximum is 80; lower values consider better outcome.
Time Frame: baseline to post-treatment (on average 24 weeks)
Population: Intention-to-Treat
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Stepped Care Program: stepped-care program with self-help module with minimal therapist contact as first step, followed by therapist-guided intervention depending on status of remission (8 sessions up to 24 sessions)
- Standardtherapy: standard therapy (therapist-guided intervention only; 16 sessions)
Arm/Group | Stepped Care Program | Standardtherapy
Number analyzed (Participants) | 46 | 43
units on a scale
  baseline | 43.13 (14.26) | 48.94 (11.00)
  post-treatment | 34.85 (14.86) | 33.35 (16.90)
Statistical Analysis 1: Comparison: Stepped Care Program vs Standardtherapy; Test type: Superiority or Other; p < 0.05, ANOVA — priori threshold for statistical significance is 0.05 p-value is not adjusted for multiple comparisons; We report the interaction effect; Mean Difference (Final Values) = 5.82 — The reported interaction effect is significant (p< .05) in favour of standard therapy

2. Secondary Outcome: Change From Baseline in Brief Symptom Inventory (BSI)
Description: The scale measures general psychopathology on 53 items on a 5-point scale (range of scores is 0-4). Minimum for all 53 items is 0, maximum is 212. Lower scores consider better outcome.
Time Frame: baseline to post-treatment (on average 24 weeks)
Population: Intention-to-Treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stepped Care Program | Standardtherapy
Number analyzed (Participants) | 46 | 43
units on a scale
  baseline | 1.00 (0.59) | 0.90 (0.56)
  post-treatment | 0.71 (0.51) | 0.51 (0.51)
Statistical Analysis 1: Comparison: Stepped Care Program vs Standardtherapy; Test type: Superiority or Other; p < 0.05, ANOVA — priori threshold for statistical significance is 0.05 p-value ist not adjusted for multiple comparisons; we report the interaction effect; Mean Difference (Final Values) = 1.24 — The reported interaction effect is not significant

3. Secondary Outcome: Change on Baseline in Center for Epidemiologic Studies Depression Scale (CES-D)
Description: The scale measures depressive symptoms on 20 items on a 4-point scale (range of scores is 0-3; minimum for all 20 items is 0, maximum 60). Lower scores consider better outcome.
Time Frame: baseline to post-treatment (on average 24 weeks)
Population: Intention-to-Treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stepped Care Program | Standardtherapy
Number analyzed (Participants) | 46 | 43
units on a scale
  baseline | 21.48 (9.97) | 21.47 (11.04)
  post-treatment | 16.20 (10.26) | 14.28 (9.93)
Statistical Analysis 1: Comparison: Stepped Care Program vs Standardtherapy; Test type: Superiority or Other; p < 0.05, ANOVA — p-value is not adjusted for multiple comparisons; we report the interaction effect; Mean Difference (Final Values) = 0.99 — The reported interaction effect is not significant

4. Primary Outcome: Change From Baseline in Social Phobia Scale (SPS)
Description: The scale measures social anxiety on a 5-point scale (range of score is 0-4) ; the number of items is 20; the total minimum for all 20 items is 0 and the total maximum is 80; lower values consider better outcome.
Time Frame: baseline to post-treatment (on average 24 weeks)
Population: Intention-to-Treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stepped Care Program | Standardtherapy
Number analyzed (Participants) | 46 | 43
units on a scale
  baseline | 35.85 (14.97) | 33.95 (13.12)
  post-treatment | 24.89 (17.41) | 17.58 (13.36)
Statistical Analysis 1: Comparison: Stepped Care Program vs Standardtherapy; Test type: Superiority or Other; p < 0.05, ANOVA — priori threshold for statistical significance is 0.05 p-value ist not adjusted for multiple comparisons; we report the interaction effect; Mean Difference (Final Values) = 3.43 — The reported interaction is not significant

5. Primary Outcome: Change From Baseline in Liebowitz Social Anxiety Scale (LSAS)
Description: The scale measures social anxiety and avoidance on a 4-point-scale (range of scores is 0-3). Blinded raters assessed social anxiety and avoidance behaviour relating to 24 social situations. Minimum for all 24 situations is 0, maximum for all 24 situations including the assessments for anxiety and avoidance is 144). Lower scores consider better outcome.
Time Frame: baseline to post-treatment (on average 24 weeks)
Population: Intention-to-Treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stepped Care Program | Standardtherapy
Number analyzed (Participants) | 46 | 43
units on a scale
  baseline | 57.46 (23.61) | 60.58 (19.37)
  post-treatment | 41.22 (23.49) | 31.84 (21.57)
Statistical Analysis 1: Comparison: Stepped Care Program vs Standardtherapy; Test type: Superiority or Other; p < 0.05, ANOVA — priori threshold for statistical significance ist 0.05 p-value ist nor adjusted for multiple comparisons; we report the interaction effect; Mean Difference (Final Values) = 6.86 — The reported interaction effect is significant (p < .05) in favour of standard therapy

ADVERSE EVENTS:
Description: No serious and/or other adverse events were assessed.
Arm/Group | Stepped Care Program | Standardtherapy
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes